CLINICAL TRIAL: NCT01102322
Title: Factors Associated With the Use of Lung Protective Ventilation Strategy (LPV) in ALI/ARDS Patients in ICU
Brief Title: Factors Associated With the Use of Lung Protective Ventilation Strategy (LPV) in Acute Lung Injury/Acute Respiratory Distress Syndrome (ALI/ARDS) Patients in Intensive Care Unit (ICU)
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jih-Shuin Jerng, Medical department of National Taiwan University Hospital
Other Study IDs: 201002021R
Record Dates: First submitted 2010-03-17; First posted 2010-04-13 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Behavioral: Quality

INTERVENTIONS:
Behavioral: Quality — Factors associated with the use of lung protective ventilation strategy (LPV) in ALI/ARDS patients in ICU

SUMMARY:
In 1967, Ashbaugh et al first described 12 patients with a syndrome characterized by the acute onset dyspnea, severe hypoxemia, diffuse lung infiltrates on the chest radiography and decreased lung compliance. Moreover, in 1988, Murray et al proposed a lung injury scoring system based on the level of positive end-expiratory pressure (PEEP), PaO2-to-FiO2 ratio, static lung compliance, degree of infiltrates on the chest radiograph, and clinical cause. A score of 2.5 or greater was considered to be consistent with a diagnosis of ARDS. The current definition of ARDS was proposed by Bernard et al and the American-European Consensus Conference in 1994. The criteria of ARDS included: 1) acute onset; 2) a PaO2/FIO2 ratio, or hypoxia score, of < 200, regardless of positive endexpiratory pressure; 3) bilateral infiltrates on chest radiograph; and 4) a pulmonary artery occlusion pressure of <18 mm Hg or the absence of clinical evidence of left atrial hypertension.

However, despite advances in ventilator management, the mortality rate of acute lung injury and the acute respiratory distress syndrome remains very high (approximately 40 to 50 percent). In 2000, ARDS Network trial compared the effects of 6 versus 12 mL/kg of tidal volume per predicted body weight (PBW) among 861 patients and noted an overall 22% reduction in mortality rate, more ventilator-free days, and more organ-failure-free days in the low-tidal-volume group. Therefore, the current approach to mechanical ventilation of a patient with ARDS emphasizes the use of lower tidal volumes with lower pressures to avoid causing lung overdistension and ventilator associated lung injury.

Nevertheless, one year after publication of the ARDSnet trial, Rubenfeld et al noted that lung-protective ventilation strategies were applied in less than 5% of patients with ARDS or ALI at a single ARDSnet center. Rubenfeld et al found that common barriers to the initiation of low tidal volume ventilation include unwillingness to relinquish control of the ventilator, failure to recognize patients as having ALI/ARDS, and perceived contraindications to low tidal volume ventilation. Significant barriers to the continuation of low tidal volume ventilation include concerns regarding patient discomfort and tachypnea or hypercapnia and acidosis.

In addition, Kalhan et al also evaluated factors associated with the choice of tidal volume and he reported that underuse of LPV may be related to clinicians' under-recognition of less severe cases of ALI, and their reserving of low-tidal volume ventilation for more severe cases, or both. However, the factors such as comorbidity and pathophysiological change associated with underuse of lung protective ventilation strategy are not clear. The investigators perform a prospective single-center study to investigate the factors associated with the use of lung protective ventilation strategy (LPV) in ALI/ARDS patients in ICU.

DETAILED DESCRIPTION:
In 1967, Ashbaugh et al first described 12 patients with a syndrome characterized by the acute onset dyspnea, severe hypoxemia, diffuse lung infiltrates on the chest radiography and decreased lung compliance. The syndrome, initially called acute respiratory distress in adult and is now named as the acute respiratory distress syndrome (ARDS). Moreover, in 1988, Murray et al proposed a lung injury scoring system based on the level of positive end-expiratory pressure (PEEP),PaO2-to-FiO2 ratio, static lung compliance, degree of infiltrates on the chest radiograph, and clinical cause. A score of 2.5 or greater was considered to be consistent with a diagnosis of ARDS. The current definition of ARDS was proposed by Bernard et al and the American-European Consensus Conference in 1994. The criteria of ARDS included: 1) acute onset; 2) a PaO2/FIO2 ratio, or hypoxia score, of <200, regardless of positive endexpiratory pressure; 3) bilateral infiltrates on chest radiograph; and 4) a pulmonary artery occlusion pressure of <18 mm Hg or the absence of clinical evidence of left atrial hypertension.

However, despite advances in ventilator management, the mortality rate of acute lung injury and the acute respiratory distress syndrome remains very high (approximately 40 to 50 percent). In 2000, ARDS Network trial compared the effects of 6 versus 12 mL/kg of tidal volume per predicted body weight(PBW) among 861 patients and noted an overall 22% reduction in mortality rate, more ventilator-free days, and more organ-failure-free days in the low-tidal-volume group. Therefore, the current approach to mechanical ventilation of a patient with ARDS emphasizes the use of lower tidal volumes with lower pressures to avoid causing lung overdistension and ventilator associated lung injury.

Nevertheless, one year after publication of the ARDSnet trial, Rubenfeld et al noted that lung-protective ventilation strategies were applied in less than 5% of patients with ARDS or ALI at a single ARDSnet center. Rubenfeld et al found that common barriers to the initiation of low tidal volume ventilation include unwillingness to relinquish control of the ventilator, failure to recognize patients as having ALI/ARDS, and perceived contraindications to low tidal volume ventilation. Significant barriers to the continuation of low tidal volume ventilation include concerns regarding patient discomfort and tachypnea or hypercapnia and acidosis.

In addition, Kalhan et al also evaluated factors associated with the choice of tidal volume and he reported that underuse of LPV may be related to clinicians' under-recognition of less severe cases of ALI, and their reserving of low-tidal volume ventilation for more severe cases, or both. However, the factors such as comorbidity and pathophysiological change associated with underuse of lung protective ventilation strategy are not clear. We perform a prospective single-center study to investigate the factors associated with the use of lung protective ventilation strategy (LPV) in ALI/ARDS patients in ICU

ELIGIBILITY:
Inclusion Criteria:

* All intubated and mechanically ventilated patients who meet the criteria of American-European Consensus Conference (AECC) criteria for ALI/ ARDS:
* Acute onset of illness
* Bilateral (patchy, diffuse, or homogeneous) infiltrates consistent with pulmonary edema
* PaO2/FiO2 <=300 (corrected for altitude): (P/F <300 for ALI and P/F <200 for ARDS)
* No clinical evidence of left atrial hypertension

Exclusion Criteria:

* Age <18 years
* Enrolled in other clinical trials
* Had confirmed alternative diagnoses that would have different clinical course than ARDS/ALI, e.g., diffuse alveolar hemorrhage, vasculitis, interstitial pneumonitis, etc.
* Congestive heart failure related pulmonary edema
* Acute myocardial infarction
* Pregnancy
* Patients with definite contraindication to the use of low-tidal volume ventilation, e.g., increased intracranial pressure, tricyclic antidepressant overdose, etc.
* The patient who meets inclusion criteria initially but rapidly improved within 24 hours of diagnosis of ARDS/ALI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute respiratory distress syndrome patients
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The rate of appropriately use of Lung Protective strategy in ALI/ARDS patients | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Shuin Jerng, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Jih-Shuin Jerng, Taipei, Taiwan